CLINICAL TRIAL: NCT03368547
Title: 68Ga-PSMA-11 PET/CT for Staging of Intermediate and High Risk Prostate Cancer Prior to Radical Prostatectomy
Brief Title: 68Ga-PSMA-11 PET/CT in Imaging Patients With Intermediate or High Risk Prostate Cancer Before Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-001684; NCI-2016-01768 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-11-27; First posted 2017-12-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2021-07

CONDITIONS: Prostate Adenocarcinoma; Stage IIB Prostate Cancer AJCC v7; Stage III Prostate Cancer AJCC v7; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (68Ga-PSMA-11, PET/CT) (Experimental): Patients receive 68Ga-PSMA-11 IV and undergo PET/CT scan over 20-50 minutes on day 1.
  Interventions: Procedure: Computed Tomography; Radiation: Gallium Ga 68 Gozetotide; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies how well 68Ga-PSMA-11 positron emission tomography (PET)/computed tomography (CT) works in imaging patients with intermediate or high risk prostate cancer before surgery. Diagnostic procedures, such as PET/CT scans, may help find and diagnose prostate cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the sensitivity and specificity of gallium Ga 68 gozetotide (68Ga-PSMA-11) PET for the detection of regional nodal metastases compared to pathology at radical prostatectomy on a per patient basis, and on a per patient basis using nodal regional correlation.

SECONDARY OBJECTIVES:

I. To assess the positive and negative predictive value of 68Ga-PSMA-11 PET for the detection of regional nodal metastases compared to pathology at radical prostatectomy on a per patient basis, and on a per patient basis using nodal regional correlation.

II. To assess sensitivity, specificity, positive and negative predictive value of 68Ga- PSMA-11 PET for the detection of extra-pelvic nodal metastases, visceral metastases and osseous metastases compared to biopsy and imaging follow-up.

OUTLINE:

Patients receive 68Ga-PSMA-11 intravenously (IV) and undergo PET/CT scan over 20-50 minutes on day 1.

After completion of study, patients are followed up at 2-4 days, then at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma
* Considered for prostatectomy with lymph node dissection
* Intermediate to high-risk disease (as determined by elevated prostate specific antigen [PSA] [PSA > 10], tumor [T]-stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors)
* Able to provide written consent
* Karnofsky performance status of >= 50 (or Eastern Cooperative Oncology Group [ECOG]/World Health Organization [WHO] equivalent)

Exclusion Criteria:

* Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam
* Neoadjuvant chemotherapy or radiation therapy prior to prostatectomy including focal ablation techniques (high-intensity focused ultrasound ablation [HiFu])

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity of 68Ga-PSMA-11 positron emission tomography for the detection of regional nodal metastases compared to pathology at radical prostatectomy on a per patient basis and using nodal regional correlation | Up to 12 months
  Will be summarized by descriptive statistics.
Specificity of 68Ga-PSMA-11 positron emission tomography for the detection of regional nodal metastases compared to pathology at radical prostatectomy on a per patient basis and using nodal regional correlation | Up to 12 months
  Will be summarized by descriptive statistics.
Positive predictive value of 68Ga-PSMA-11 positron emission tomography for the detection of regional nodal metastases compared to pathology at radical prostatectomy on a per patient basis and using nodal regional correlation | Up to 12 months
  Will be summarized by descriptive statistics.
Negative predictive value of 68Ga-PSMA-11 positron emission tomography for the detection of regional nodal metastases compared to pathology at radical prostatectomy on a per patient basis and using nodal regional correlation | Up to 12 months
  Will be summarized by descriptive statistics.

SECONDARY OUTCOMES:
Sensitivity of 68Ga-PSMA-11 positron emission tomography for the detection of extra-pelvic nodal metastases, visceral metastases, and osseous metastases compared to biopsy and imaging follow-up | Up to 12 months
  Will be summarized by descriptive statistics.
Specificity of 68Ga-PSMA-11 positron emission tomography for the detection of extra-pelvic nodal metastases, visceral metastases, and osseous metastases compared to biopsy and imaging follow-up | Up to 12 months
  Will be summarized by descriptive statistics.
Positive predictive value of 68Ga-PSMA-11 positron emission tomography for the detection of extra-pelvic nodal metastases, visceral metastases, and osseous metastases compared to biopsy and imaging follow-up | Up to 12 months
  Will be summarized by descriptive statistics.
Negative predictive value of 68Ga-PSMA-11 positron emission tomography for the detection of extra-pelvic nodal metastases, visceral metastases, and osseous metastases compared to biopsy and imaging follow-up | Up to 12 months
  Will be summarized by descriptive statistics.

OTHER OUTCOMES:
Sensitivity for detection of regional nodal metastases in comparison to cross sectional imaging performed contemporaneously with the 68Ga-PSMA-11 positron emission tomography | Up to 12 months
  Will be summarized by descriptive statistics.
Specificity for detection of regional nodal metastases in comparison to cross sectional imaging performed contemporaneously with the 68Ga-PSMA-11 positron emission tomography | Up to 12 months
  Will be summarized by descriptive statistics.
Positive predictive value for detection of regional nodal metastases in comparison to cross sectional imaging performed contemporaneously with the 68Ga-PSMA-11 positron emission tomography | Up to 12 months
  Will be summarized by descriptive statistics.
Negative predictive value for detection of regional nodal metastases in comparison to cross sectional imaging performed contemporaneously with the 68Ga-PSMA-11 positron emission tomography | Up to 12 months
  Will be summarized by descriptive statistics.
PSA progression free survival | Up to 1 year
  Will compare patients with and without pelvic nodal metastases.
Standardized uptake value maximum and short axis diameter of nodal disease on cross sectional imaging correlated to presence of true pathology | Up to 12 months
Incidence of osseous and distant metastatic lesions | Up to 12 months
Impact of 68Ga-PSMA-11 positron emission tomography on clinical management | Up to 12 months
Incidence of adverse events | Up to 3 days
  Assessed per Common Terminology Criteria for Adverse Events version 4.03.
Inter-reader reproducibility | Up to 12 months
Sensitivity and specificity on lesions level for 68Ga-PSMA-11 positron emission tomography and multiparametric magnetic resonance imaging | Up to 12 months
Quantitative parameters for malignant and benign lesions (BPH, hgPIN, inflammation) in 68Ga-PSMA-11 positron emission tomography and multiparametric magnetic resonance imaging | Up to 12 months
Gross-tumor-volume using 68Ga-PSMA-11 positron emission tomography and multiparametric magnetic resonance imaging | Up to 12 months
  Will be compared to tumor extent in histopathology.
Lesional standardized uptake value maximum from 68Ga-PSMA-11 | Up to 12 months
  Will be correlated with immunohistochemical stainings (e.g. PSMA, PI3K, Akt) and Gleason score.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Djaileb L, Armstrong WR, Thompson D, Gafita A, Farolfi A, Rajagopal A, Grogan TR, Nguyen K, Benz MR, Hotta M, Barbato F, Ceci F, Schwarzenbock SM, Unterrainer M, Zacho HD, Juarez R, Cooperberg M, Carroll P, Washington S, Reiter RE, Eiber M, Herrmann K, Fendler WP, Czernin J, Hope TA, Calais J. Presurgical 68Ga-PSMA-11 Positron Emission Tomography for Biochemical Recurrence Risk Assessment: A Follow-up Analysis of a Multicenter Prospective Phase 3 Imaging Trial. Eur Urol. 2023 Dec;84(6):588-596. doi: 10.1016/j.eururo.2023.06.022. Epub 2023 Jul 21. PMID 37482512
- [Derived] Sonni I, Felker ER, Lenis AT, Sisk AE, Bahri S, Allen-Auerbach M, Armstrong WR, Suvannarerg V, Tubtawee T, Grogan T, Elashoff D, Eiber M, Raman SS, Czernin J, Reiter RE, Calais J. Head-to-Head Comparison of 68Ga-PSMA-11 PET/CT and mpMRI with a Histopathology Gold Standard in the Detection, Intraprostatic Localization, and Determination of Local Extension of Primary Prostate Cancer: Results from a Prospective Single-Center Imaging Trial. J Nucl Med. 2022 Jun;63(6):847-854. doi: 10.2967/jnumed.121.262398. Epub 2021 Oct 14. PMID 34649942
- [Derived] Hope TA, Eiber M, Armstrong WR, Juarez R, Murthy V, Lawhn-Heath C, Behr SC, Zhang L, Barbato F, Ceci F, Farolfi A, Schwarzenbock SM, Unterrainer M, Zacho HD, Nguyen HG, Cooperberg MR, Carroll PR, Reiter RE, Holden S, Herrmann K, Zhu S, Fendler WP, Czernin J, Calais J. Diagnostic Accuracy of 68Ga-PSMA-11 PET for Pelvic Nodal Metastasis Detection Prior to Radical Prostatectomy and Pelvic Lymph Node Dissection: A Multicenter Prospective Phase 3 Imaging Trial. JAMA Oncol. 2021 Nov 1;7(11):1635-1642. doi: 10.1001/jamaoncol.2021.3771. PMID 34529005
- [Derived] Ma TM, Gafita A, Shabsovich D, Juarez J, Grogan TR, Thin P, Armstrong W, Sonni I, Nguyen K, Lok V, Reiter RE, Rettig MB, Steinberg ML, Kupelian PA, Yang DD, Muralidhar V, Chu C, Feng F, Savjani R, Deng J, Parikh NR, Nickols NG, Elashoff D, Czernin J, Calais J, Kishan AU. Identifying the Best Candidates for Prostate-specific Membrane Antigen Positron Emission Tomography/Computed Tomography as the Primary Staging Approach Among Men with High-risk Prostate Cancer and Negative Conventional Imaging. Eur Urol Oncol. 2022 Feb;5(1):100-103. doi: 10.1016/j.euo.2021.01.006. Epub 2021 Feb 16. PMID 33602654
- [Derived] Lenis AT, Pooli A, Lec PM, Sadun TY, Johnson DC, Lebacle C, Fendler WP, Eiber M, Czernin J, Reiter RE, Calais J. Prostate-specific Membrane Antigen Positron Emission Tomography/Computed Tomography Compared with Conventional Imaging for Initial Staging of Treatment-naive Intermediate- and High-risk Prostate Cancer: A Retrospective Single-center Study. Eur Urol Oncol. 2022 Oct;5(5):544-552. doi: 10.1016/j.euo.2020.08.012. Epub 2020 Sep 18. PMID 32958451